CLINICAL TRIAL: NCT00409071
Title: Placebo-controlled Evaluation of Homeopathic Remedy (Cocculine®) Efficacy in the Management of Nausea After Adjuvant Chemotherapy in Non Metastatic Breast Cancer.
Brief Title: Placebo-controlled Evaluation of Cocculine® Efficacy in the Management of Nausea After Chemotherapy in Breast Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: BOIRON (Industry)
Responsible Party: Zora ABDELBOST, Research Direction
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COCCULINE; ET2005-028
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-02

CONDITIONS: Breast Cancer
Keywords: Non metastatic breast cancer; Adjuvant chemotherapy; Nausea; Vomiting; Quality of life; Homeopathy
MeSH Terms: conditions — Breast Neoplasms; Nausea; Vomiting | interventions — sinomenine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): cocculine
  Interventions: Drug: Cocculine®
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Cocculine® — 12 tablets in 3 days at each of the CT courses: 2 on the day before evening of the CT courses; 2 on the morning, noon and evening of the CT courses; 2 on morning and noon of the day after the CT courses.
  Arms: 1
Drug: placebo — 12 tablets in 3 days at each of the CT courses: 2 on the day before evening of the CT courses; 2 on the morning, noon and evening of the CT courses; 2 on morning and noon of the day after the CT courses.
  Arms: 2

SUMMARY:
The purpose of the study is to determine whether a homeopathic remedy (Cocculine®) is effective in the prevention of chemotherapy-induced nausea in non metastatic breast cancer.

Eligible patients will be randomly assigned to one of 2-arms: Cocculine® or placebo.

The number of patients required to demonstrate a 0.5-point reduction in nausea on a visual analogue scale, assuming an alpha risk of 5% in a two-sided test and 85% power, is 396 (198 per arm). It has been estimated that the enrollment period should be 18 months.

DETAILED DESCRIPTION:
The proportion of women with breast cancer treated by chemotherapy (CT) is increasing. CT-induced nausea and vomiting negatively impact patient quality of life.

The primary objective of the trial is to evaluate against a placebo the efficacy of Cocculine® administered as an adjunct to conventional treatments (corticosteroids and 5-HT3 receptor antagonists) for the management of nausea induced by a 1st course of adjuvant CT with FAC50, FEC100 or TAC in patients with non-metastatic breast cancer.

Secondary objectives are to test:

* the persistence of Cocculine® efficacy over the 2nd and 3rd CT courses
* the contribution of Cocculine® to the global management of nausea and vomiting during adjuvant CT
* patient compliance with Cocculine® dose.

Eligible patients will be randomly assigned to one of 2 arms: Cocculine® or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically proven non metastatic breast cancer
* No previous chemotherapy
* Treatment planning including 6 adjuvant CT courses with the first 3 being necessarily of the FAC50, FEC100 or TAC type
* Age>= 18 years
* ECOG performance status (PS) <= 2 (WHO scale)
* Patient able to read and understand French
* Written, voluntary, informed consent

Exclusion Criteria:

* Previous treatment with chemotherapy (including neo-adjuvant chemotherapy for breast cancer)
* Previous malignancies (except basal cell skin cancer or cervical cancer in situ or any other curatively treated malignancy in complete remission for more than 5 years)
* Contraindication to corticosteroids or 5-HT3 receptor antagonists
* Treatment with Cocculine® or any other anti-emetic drug in the 15 days before inclusion
* Pregnant or lactating women
* Follow-up impossible for social, geographical, familial or psychological reasons
* Patients who cannot be contacted by phone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2005-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Score of "nausea" calculated using the FLIE questionnaire (Functional Living index for Emesis with 5-day recall)at the time of the 1rst adjuvant CT course | The nausea items of FLIE questionnaire are completed by patients on the 6th day of the 1st course.

SECONDARY OUTCOMES:
Score of "vomiting" and global score of "nausea + vomiting" calculated using the FLIE questionnaire at the time of the 1st, 2nd and 3rd adjuvant CT courses | Nausea and vomiting items of FLIE questionnaire are completed by patients on the 6th day of the 1st, 2nd and 3rd adjuvant CT courses
Score of "nausea" calculated using the FLIE questionnaire at the time of the 2nd and 3rd adjuvant CT courses | Nausea items of FLIE questionnaire are completed by patients on the 6th day of the 2nd and 3rd adjuvant CT courses
Patient autoevaluation (D1-D5) of nausea severity using a visual analogue scale and of the frequency of vomiting during the 1st, 2nd and 3rd adjuvant CT courses | Visual analogue scale are completed by patients the 1st five days of the 1st, 2nd and 3rd adjuvant CT courses
Rate of toxic effects (nausea and vomiting) recorded by investigators at the end of each of the 6 CT courses | Recorded by investigators at the end of each of the 6 CT courses
Evaluation of compliance: patient autoevaluation and counting of remaining tablets | Patients register date and hour of tablets taking on a diary. Box remaining tablets will be count at the end of the 6 CT courses.

CONTACTS AND LOCATIONS:
Overall Officials: RAY-COQUARD Isabelle, MD, Principal Investigator — Centre Leon Berard, France
Locations (1):
- Centre Leon Berard, Lyon, France

REFERENCES:
- [Background] Pommier P, Gomez F, Sunyach MP, D'Hombres A, Carrie C, Montbarbon X. Phase III randomized trial of Calendula officinalis compared with trolamine for the prevention of acute dermatitis during irradiation for breast cancer. J Clin Oncol. 2004 Apr 15;22(8):1447-53. doi: 10.1200/JCO.2004.07.063. PMID 15084618
- [Derived] Perol D, Provencal J, Hardy-Bessard AC, Coeffic D, Jacquin JP, Agostini C, Bachelot T, Guastalla JP, Pivot X, Martin JP, Bajard A, Ray-Coquard I. Can treatment with Cocculine improve the control of chemotherapy-induced emesis in early breast cancer patients? A randomized, multi-centered, double-blind, placebo-controlled Phase III trial. BMC Cancer. 2012 Dec 17;12:603. doi: 10.1186/1471-2407-12-603. PMID 23244208